CLINICAL TRIAL: NCT04477603
Title: Use of the Impella ECP in Patients Undergoing an Elective or Urgent High-Risk Percutaneous Coronary Intervention: An Early Feasibility Study
Brief Title: Impella ECP Early Feasibility Study
Acronym: ECP EFS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: TMF-VV-17471
Record Dates: First submitted 2020-07-13; First posted 2020-07-20 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-07

CONDITIONS: High-risk Percutaneous Coronary Intervention
Keywords: HRPCI; High-risk percutaneous coronary intervention; circulatory support; left ventricular unloading; Abiomed; Impella; Impella ECP

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Subjects receiving the Impella ECP (Experimental)
  Interventions: Device: Impella ECP

INTERVENTIONS:
Device: Impella ECP — Subjects will receive the Impella ECP prior to high-risk percutaneous intervention. Device escalation or early termination of the study will be allowed for subjects as deemed necessary by the treating physician. Subjects will be followed until 30-days post-intervention.

SUMMARY:
The Impella ECP EFS is a prospective, multicenter, single-arm, feasibility study evaluating the safety of the Impella ECP device in adult patients undergoing an elective or urgent high-risk percutaneous coronary intervention.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-arm, feasibility study evaluating the safety of the Impella ECP device in adult patients undergoing an elective or urgent high-risk percutaneous coronary intervention (HRPCI). Additionally, this study will evaluate the feasibility of placing the ECP pump across the aortic valve without the use of a guidewire and assess the ability of the pump to provide sufficient hemodynamic support during a HRPCI. Investigational device products include: Impella ECP pump system (a percutaneous transvalvular micro-axial blood pump), 9Fr introducer sheath, and the automated Impella controller with revised console software to allow control of the Impella ECP.

Following informed consent, subjects eligible for a HRPCI that meet all of the inclusion and none of the exclusion criteria will be enrolled into the study. The intended coronary intervention is then carried out under mechanical circulatory support by the Investigational Device. This device is inserted through a sheath that has been deployed through a femoral puncture, following crimping of the Impella ECP. After proper placement and wireless passage of the aortic valve, the device pumps blood from the left ventricle into the aorta. Once the interventional procedure is completed, the device is weaned and removed. Subjects will be followed up until 30 days post intervention.

The primary and secondary end points will be summarized and presented without formal statistical testing. Safety will be assessed by the rate of composite Major Device-Related Adverse Events, evaluated at the end of the HRPCI procedure. Feasibility is defined as the successful delivery, initiation and maintenance of sufficient hemodynamic support to increase in or maintenance the MAP at physiologic levels (> 60 mmHg), evaluated up to the end of procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 90 years
2. Subject has signed the informed consent
3. Scheduled for an elective or urgent high risk percutaneous coronary intervention with hemodynamic support

Exclusion Criteria:

1. Aortic valve disease that is anticipated to be prohibitive to Impella ECP crossing, including greater than mild aortic stenosis
2. Previous aortic valve replacement or reconstruction
3. Thrombus in left ventricle
4. Subjects with known aortic vessel disease or with aortic dissection
5. Any contraindication that precludes placing an Impella including aortic, iliac or femoral disease such as tortuosity, extensive atherosclerotic disease or stenosis
6. Prior stroke with any permanent neurologic deficit or any prior intracranial hemorrhage or any prior subdural hematoma or known intracranial pathology pre-disposing to intracranial bleeding, such as an arteriovenous malformation or mass
7. Cardiogenic shock or acutely decompensated pre-existing chronic heart failure. Cardiogenic shock is defined as: systemic hypotension (systolic BP <90 mmHg or the need for inotropes/pressors to maintain a systolic BP >90 mmHg) plus one of the following: any requirement for pressors/inotropes prior to arrival at the catheterization laboratory, clinical evidence of end-organ hypoperfusion or use of IABP or any other circulatory support device
8. Infection of the proposed procedural access site or suspected systemic active infection, including any fever
9. Subject has previously been symptomatic with or hospitalized for COVID-19 unless he/she has been discharged (if hospitalized) and asymptomatic for ≥8 weeks and has returned to his/her prior baseline (pre-COVID) clinical condition
10. Known contraindication to heparin (i.e., heparin-induced thrombocytopenia), contrast media or Study-required medication(s) (i.e., aspirin)
11. Platelet count <75k, bleeding diathesis, coagulopathy or unwilling to receive blood transfusions
12. Subject is on dialysis
13. Suspected or known pregnancy
14. Subject has other medical, social or psychological problems that, in the opinion of the Investigator, compromises the subject's ability to give written informed consent and/or to comply with study procedures
15. Participation in the active treatment or follow-up phase of another clinical study of an investigational drug or device which has not reached its primary endpoint
16. Subject belongs to a vulnerable population [Vulnerable subject populations are defined as individuals with mental disability, persons in nursing homes, children, impoverished persons, homeless persons, nomads, refugees and those permanently incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces and persons kept in detention]

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-09 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility: successful hemodynamic support | through end of procedure, 1 day
  The feasibility assessment is defined as the successful delivery, initiation and maintenance of sufficient hemodynamic support to increase in or maintenance the MAP at physiologic levels (> 60 mmHg)
Safety: Major Device-Related Adverse Events | through end of procedure, 1 day
  The rate of composite Major Device-Related Adverse Events

SECONDARY OUTCOMES:
Technical Success | through end of procedure, 1 day
  The ability to complete the entire Impella ECP delivery procedure and pump initiation without device malfunction.
Procedural Success | through end of procedure, 1 day
  Technical success with a sufficient flow generation by the pump in order to increase or maintain MAP during the interventional procedure.
Rate of each individual Major Device-Related Adverse Event | through end of study, 30 days
  The rate of each individual Major Device-Related Adverse Event.
Rate of composite Major Device-Related Adverse Events | through end of study, 30 days
  The rate of composite Major Device-Related Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Kaki, MD, Principal Investigator — Ascension St. John Hospital; Seth Bilazarian, MD, Study Director — Abiomed Inc.; Navin Kapur, MD, Study Director — Abiomed Inc.
Locations (5):
- United States (5):
  - Tufts Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health St. John Hospital, Detroit, Michigan
  - The Valley Hospital, Paramus, New Jersey
  - The Christ Hospital, Cincinnati, Ohio